CLINICAL TRIAL: NCT06946160
Title: A Phase I/III, Randomized, Two-armed, Double-blinded, Parallel, Active-controlled, Non-inferiority Clinical Trial to Compare Efficacy and Safety of AbobotulinumtoxinA (Espad Pharmed) Versus AbobotulinumtoxinA (Dysport®, Ipsen Co.) for Correction of Moderate to Severe Glabellar Lines
Brief Title: A Non-inferiority Clinical Trial to Compare Efficacy and Safety of Abobotulinumtoxin A (Espad Pharmed) Versus AbobotulinumtoxinA (Dysport®, Ipsen Co.) for Correction of Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Espad Pharmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BOT.ESP.AF.III.02; IRCT20150101020514N23 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Glabellar Lines; Glabellar Frown Lines
Keywords: glabellar lines; AbobotulinumtoxinA
MeSH Terms: interventions — abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abobotulinumtoxin A (produced by Espad Pharmed Darou Co.) (Experimental): Vial of AbobotulinumtoxinA (produced by Espad Pharmed Darou Co.), administered via deep intramuscular injection into 3 to 5 sites in the glabellar area using a 1 ml syringe, with a total dose of 40 to 60 International Units (IU), administered in a single treatment session.
  Interventions: Drug: Abobotulinumtoxin A (Espad Pharmed Darou Co.)
- Abobotulinumtoxin A (Dysport®, produced by Ipsen Co.) (Active Comparator): Vial of AbobotulinumtoxinA (Dysport®, produced by Ipsen Co.), administered via deep intramuscular injection into 3 to 5 sites in the glabellar area using a 1 ml syringe, with a total dose of 40 to 60 International Units (IU), administered in a single treatment session.
  Interventions: Drug: Abobotulinumtoxin A (Ipsen Co.)

INTERVENTIONS:
Drug: Abobotulinumtoxin A (Espad Pharmed Darou Co.) — Vial of Abobotulinumtoxin A (produced by Espad Pharmed Darou Co.), administered via deep intramuscular injection
  Arms: Abobotulinumtoxin A (produced by Espad Pharmed Darou Co.)
Drug: Abobotulinumtoxin A (Ipsen Co.) — Vial of AbobotulinumtoxinA (Dysport®, produced by Ipsen Co.), administered via deep intramuscular injection
  Arms: Abobotulinumtoxin A (Dysport®, produced by Ipsen Co.)

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of AbobotulinumtoxinA (produced by Espad Pharmed Darou Co.) for correction of moderate to severe glabellar lines.

Hypothesis: AbobotulinumtoxinA (produced by Espad Pharmed Darou Co.) has acceptable efficacy and safety profile for correction of moderate to severe glabellar lines.

Primary Outcome: To verify the non-inferiority of the efficacy of AbobotulinumtoxinA (produced by Espad Pharmed Darou Co.) compared with AbobotulinumtoxinA (Dysport®, produced by Ipsen Co.) by percentage of responders at maximum frown at day 30 after treatment.

Researchers will compare the efficacy and safety profile of AbobotulinumtoxinA (produced by Espad Pharmed Darou Co.) with AbobotulinumtoxinA (Dysport®, produced by Ipsen Co.).

The study is designed as phase III, randomized, two armed, double-blind, parallel, active controlled, non-inferiority clinical trial.

Participants received a total dose of 40-60 units into 3 to 5 sites. After two weeks, a touch-up intervention could be done based on physician's assessment.

DETAILED DESCRIPTION:
The study schedule includes Visit 0 (Screening), Visit 1 (Intervention, Day 0), and Follow-up Visits 2 (Day 14), 3 (Day 30), 4 (Day 90), and 5 (Day 120). At Visit 0, informed consent is obtained, and eligibility is assessed through initial evaluations and review of inclusion and exclusion criteria. At Visit 1, subjects are randomized (1:1) and receive the investigational treatment. Full-face photographs are obtained at Visit 1 (Before receiving the investigational treatment), and at Follow-up Visits 2, 3, 4, and 5, in both resting state and maximum frown. Efficacy is evaluated at Visits 3, 4, and 5. All adverse events are Recorded at all visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 to ≤65 years of age
2. Willingness for signing and having signed the informed consent form
3. Moderate to severe glabellar wrinkle at maximum frown based on glabellar lines severity scale (GLSS)
4. be able to participate in the visit schedules and the study procedures.

Exclusion Criteria:

1. Hypersensitivity to botulinum toxin or any other component of the formulation, as well as to injectable fillers in the facial region.
2. Previous treatment with botulinum toxin in facial areas within the past 6 months.
3. Previous treatment with dermal fillers, dermabrasion, or photo rejuvenation in the glabellar region within the past 12 months.
4. History of dermal filler injection in the forehead region within the past year.
5. History of eyebrow tattooing or any other procedure involving the eyebrow area within the past month.
6. Use of aminoglycosides, penicillamine, quinine, chloroquine, hydroxychloroquine, or calcium channel blockers within the past week.
7. Use of anticoagulants or aspirin within the past 10 days (participants are not required to discontinue their anticoagulant therapy to be enrolled in the study).
8. History of any cosmetic surgery (e.g., filler injections, chemical peels, or laser treatments) or use of products that induce skin remodeling or significantly affect the forehead area or its surroundings, including any aesthetic procedure involving the glabellar lines within the past 6 months.
9. History of any surgical procedure involving facial muscles or scarring in the forehead or surrounding areas (including the eyebrows).
10. Any planned aesthetic procedure involving the upper face during the course of the study.
11. Presence of disorders that may affect neuromuscular function (e.g., myasthenia gravis, amyotrophic lateral sclerosis [ALS], or Eaton-Lambert syndrome).
12. History of facial nerve paralysis.
13. Presence of clearly visible and defined facial asymmetry.
14. Ptosis of the eyelids or eyebrows due to facial muscle paralysis or a history thereof.
15. Presence of any active infection or acute dermatological condition in the injection areas.
16. Pregnancy (confirmed by urine test) or lactation.
17. Participation in other clinical studies within 30 days prior to randomization or intention to participate in other clinical trials.
18. Any other condition or circumstance that may pose a risk to the participant or interfere with the satisfactory completion of the clinical outcome.
19. History of participation in other clinical trials involving botulinum neurotoxin products or fillers within the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Responders at maximum frown by investigator's assessment | Day 30
  Percentage of responders measured by the investigator's live assessment based on Glabellar Line Severity Scale (GLSS) at maximum frown at day 30 after treatment The Glabellar Line Severity Scale (GLSS) is a 4-grade scale defined as follows: 0 = no glabellar lines, 1 = mild lines, 2 = moderate lines, 3 = severe lines. Higher scores indicate more severe glabellar lines. Participants were considered responders if they showed a reduction of at least 2 points from baseline on the scale.

SECONDARY OUTCOMES:
Responders at rest by investigator's assessment | Days 30, 90 and 120
  Percentage of responders measured by the investigator's live assessment based on Glabellar Line Severity Scale (GLSS) at rest at days 30, 90 and 120 after treatment The Glabellar Line Severity Scale (GLSS) is a 4-grade scale defined as follows: 0 = no glabellar lines, 1 = mild lines, 2 = moderate lines, 3 = severe lines. Higher scores indicate more severe glabellar lines. Participants were considered responders if they showed a reduction of at least 2 points from baseline on the scale.
Responders at maximum frown by subject's self-assessment | days 30, 90 and 120
  Percentage of responders measured by the subject's self-assessment (SSA) at maximum frown at days 30, 90 and 120 after treatment The 4-grade subject's self-assessment scale defined as follows: 0 = no glabellar lines, 1 = mild lines, 2 = moderate lines, 3 = severe lines. Higher scores indicate more severe glabellar lines. Responders are defined as those reporting a reduction of at least 2 points from baseline.
Responders at rest by subject's self-assessment | days 30, 90 and 120
  Percentage of responders measured by the subject's self-assessment (SSA) at rest at days 30, 90 and 120 after treatment The 4-grade subject's self-assessment scale defined as follows: 0 = no glabellar lines, 1 = mild lines, 2 = moderate lines, 3 = severe lines. Higher scores indicate more severe glabellar lines. Responders are defined as those reporting a reduction of at least 2 points from baseline.
Responders at maximum frown by investigator's assessment | days 90 and 120
  Percentage of responders measured by the investigator's live assessment based on Glabellar Line Severity Scale (GLSS) at maximum frown at days 90 and 120 after treatment The Glabellar Line Severity Scale (GLSS) is a 4-grade scale defined as follows: 0 = no glabellar lines, 1 = mild lines, 2 = moderate lines, 3 = severe lines. Higher scores indicate more severe glabellar lines. Participants were considered responders if they showed a reduction of at least 2 points from baseline on the scale.
Total injected dose (visit 1 and touch-up visit) | Day 14
Onset of action measured by the subject's self-assessment (SSA) at rest | Day 14
  The participants were asked to record the date on which they first noticed the onset of the product's efficacy and to inform the investigator of this date during the visit on day 14.
Onset of action measured by the subject's self-assessment (SSA) at maximum frown | Day 14
  The participants were asked to record the date on which they first noticed the onset of the product's efficacy and to inform the investigator of this date during the visit on day 14.
Safety assessment by evaluation of adverse events (AEs) | Visit 0 (screening), visit 1 (Day 0), visit 2 (Day 14), visit 3 (Day 30), visit 4 (Day 90), visit 5 (Day 120)
  Adverse events (AEs) were assessed at all visits. All reported events were classified as mild, moderate, or severe. Moreover, seriousness of Adverse events was assessed according to International Council for Harmonization (ICH-E2B) guidelines. The causality relation was assessed based on the World Health Organization (WHO) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Firooz, Medical Doctor, Principal Investigator — Center for Research and Training in Skin Diseases and Leprosy, Tehran, Tehran 1416613675
Locations (1):
- Center for Research and Training in Skin Diseases And Leprosy, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No
Data produced in the present study are available upon reasonable request from the investigators.